CLINICAL TRIAL: NCT00827801
Title: MDASI-HF: Bridging the Symptom Management Gap in Patients With Cancer and Concurrent Heart Failure to Improve Outcomes
Brief Title: M. D. Anderson Symptom Inventory - Heart Failure (MDASI-HF) Symptom Management Program
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-0722
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Heart Failure; Cancer
Keywords: Cancer; Heart Failure; HF; Cancer and Concurrent Heart Failure; MDASI-HF Symptom Management Program; MDASI-HF; MDASI-HF questionnaire; M. D. Anderson Symptom Inventory - Heart Failure; Questionnaire; Symptom Management Gap
MeSH Terms: conditions — Heart Failure; Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1: MDASI-HF questionnaire provided to Doctor for symptom management.
  Interventions: Behavioral: MDASI-HF Questionnaire
- Group 2: MDASI-HF questionnaire collected not provided to Doctor.
  Interventions: Behavioral: MDASI-HF Questionnaire

INTERVENTIONS:
Behavioral: MDASI-HF Questionnaire — M. D. Anderson Symptom Inventory - Heart Failure (MDASI-HF) questionnaire rating symptoms given in clinic Day 1, Weeks 4 & 8.
  Other Names: survey

SUMMARY:
Primary Objective:

To determine if there is a reduction in the mean symptom severity scores for the heart failure specific symptom items between baseline and at the end of three months between patients whose symptoms are managed using the MDASI-HF symptom assessment scores (treatment group) as a decision making guide, as compared to patients managed without using the MDASI-HF symptom assessment scores (control group).

Secondary Objectives:

1. Examine the correlation between mean symptom severity scores and the secondary endpoints of: a) exercise tolerance ( 6-minute walk), b) NYHA (New York Heart Association) functional classification, c) B-type natriuretic peptide (a biomarker for heart failure), and d) dose titration of HF (heart failure) medications.
2. Define symptom severity critical values in cancer patients with concurrent heart failure that trigger clinical intervention
3. Identify symptom clusters which may occur in cancer patients with concurrent heart failure.

DETAILED DESCRIPTION:
Background for Study:

Heart failure means that the heart isn't pumping as well as it should be. Your body depends on the heart's pumping action to deliver oxygen- and nutrient-rich blood to the body's cells. When the cells are nourished properly, the body can function normally. With heart failure, the weakened heart can't supply the cells with enough blood. This results in fatigue and shortness of breath. Everyday activities such as walking, climbing stairs, or carrying groceries can become very difficult.

In the standard of care, patients tell their healthcare staff about their symptoms and are treated accordingly. The MDASI-HF program is a tool that is designed to try to improve this process by measuring how severe symptoms may be in patients with cancer and heart failure, as well as measuring how these symptoms may be affecting these patients' daily lives.

To take part in the MDASI-HF program, patients complete a questionnaire at clinic visits and at home. The home questionnaire is done over the phone. The symptom information that the patients report is provided to the healthcare staff, allowing the healthcare staff to closely monitor the symptoms and respond as needed.

You must have permission from your cardiologist in order to take part in this study.

Study Groups:

If you agree to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups. However, for your safety, the doctor may assign you to a certain group based on factors such as your age, sex, and the status of the heart disease.

All participants will complete the MDASI-HF questionnaire, which asks about symptoms. If you are in Group 1, your questionnaire responses will be provided to your doctor so the doctor can use that information to manage your symptoms. If you are in Group 2, your questionnaire responses, completed either in person or via phone, will not be provided to your doctor. All participants in this study will receive appropriate medical care for management of symptoms. Both groups will have all the same procedures.

Study Visits:

During this study, you will have a clinic visit to your doctor's office on Day 1 of the study and at Weeks 4, 8, and 12.

On Day 1, the following tests and procedures will be performed:

* You will watch a patient and family education video while you wait for the doctor. The video discusses heart failure, drugs, diet, exercise, and emotional issues related to living with heart failure. The video is less than 15 minutes long.
* You will be given a patient diary and a booklet that explains how to manage heart failure. You will complete this diary once a day, which should take about 5-10 minutes each time. In this diary, you will record your weight, blood pressure, and any drugs you are taking. You should bring the diary back to the clinic at each study visit to have it reviewed.
* You will complete the MDASI-HF questionnaire in the clinic. This questionnaire asks you to rate your symptoms on a scale of 0 to 10. A score of 0 would mean the symptom is not happening and a score of 10 means the symptom is at its worst. The symptoms include heart-related symptoms and other symptoms that may be related to cancer or treatments. The questionnaire also asks you how the symptoms may have interfered with your daily life. Completing the questionnaire should take about 15 minutes.
* The distance you are able to walk in 6 minutes will be measured. You will sign a separate consent form that will describe this 6-minute walk test in more detail.
* Blood (about 1 teaspoon) will be drawn for routine tests.
* Blood (about 1 teaspoon) will be drawn for biomarker testing. The biomarker being studied is a chemical "marker" in the blood that may be related to heart failure.
* If you have not had one in the last 90 days, you will have an echocardiogram performed to check your heart function as part of your standard of care.
* If you have not had one in the last month, you will have an electrocardiogram (ECG -- a test that measures the electrical activity of the heart).

At Weeks 4 and 8, you will complete the MDASI-HF questionnaire in the clinic. Blood (about 2 teaspoons) will be drawn for routine tests. Blood (about 1 teaspoon) will be drawn for biomarker testing.

Phone Questionnaire Completion Between Visits:

Between study visits (at Weeks 1, 2, 3, 5, 6, 7, 9, 10, and 11), you will receive a phone call once a week. The phone system is "automated," and it asks you the same MDASI-HF questions as the questionnaire that you completed at the clinic. For all of the questions, you will enter a number on your phone's keypad to answer the questions. Completing the phone questionnaire should take about 10-15 minutes each time. At the end of the phone questionnaire, the system will direct you in scheduling your next call.

For Group 1 participants only, if you report that any pain or shortness of breath symptoms at 5, or any other symptom is as severe as 7 or higher, the phone system will automatically contact the clinic nurse using an alert. The nurse will call you back within 24 hours. Based on the symptom(s), the nurse will advise you about what to do next (for example, change the dose of your drugs, come in to the clinic, or go to the emergency center). The nurse will also contact your doctor right away if necessary. In addition to reviewing these severe symptoms that you may report, the study staff will be reviewing all of your questionnaire responses on a routine basis.

For Group 2 participants only, your telephone answers will not contact a clinic nurse. If you experience severe pain, shortness of breath, or your symptoms worsen, please contact the clinic nurse right away at the numbers in your instruction booklet.

Management of Symptoms:

No matter if you are in Group 1 or Group 2, if at any time you notice that any of your symptoms seem to be getting worse, you should call the clinic nurse right away at the numbers in your instruction booklet. The clinic nurse will follow up to advise you about what to do next. For example, the nurse may change the dose of your drugs, tell you to come into the clinic, or tell you to go to the emergency center. The nurse will also contact your doctor right away, if necessary.

If you feel your symptoms are severe, visit the emergency room or call 911.

End-of-Study Visit:

At Week 12, the following tests and procedures will be performed:

* You will complete the MDASI-HF questionnaire using the computer in the clinic.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* Blood (about 1 teaspoon) will be drawn for biomarker testing.
* You will perform a 6-minute walk test.
* An echocardiogram and ECG will be performed.

After the Week 12 visit, your participation in this study will be over.

This is an investigational study. At this time, the MDASI-HF program is only being used in research.

Up 144 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. All cancer patients with a concurrent diagnosis of heart failure. Heart failure can be systolic (<40% ejection fraction) or diastolic (>40% ejection fraction). Functioning at New York Heart Association class II, III, or IV.
2. Age 18 years and older
3. Able to give informed consent to participate
4. Working phone number to contact patient
5. Live within the 100 mile radius of the Houston area while enrolled in the study for the three month duration

Exclusion Criteria:

1. Younger than 18 years old
2. With a known diagnosis of dementia or Alzheimer's disease
3. Not familiar with the English language. The MDASI-HF is currently available in the English language only.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All cancer patients, 18 years of age or older, with a concurrent diagnosis of heart failure, newly diagnosed or diagnosed within past 1 year.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2009-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Mean Symptom Severity Scores (MDASI-HF Symptom Assessment Scores) | Baseline and at end of 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Anecita Fadol, PhD, MS, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org